CLINICAL TRIAL: NCT00085696
Title: A Phase 2 Study of VELCADE® (Bortezomib) With Rituximab in Subjects With Relapsed or Refractory Indolent B-Cell Lymphoma
Brief Title: VELCADE® (Bortezomib) With Rituximab in Subjects With Relapsed or Refractory Indolent B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M34103-061
Record Dates: First submitted 2004-06-11; First posted 2004-06-15 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-02

CONDITIONS: B-Cell Lymphoma; Follicular Lymphoma; Marginal Lymphoma
Keywords: Lymphoma; Non-Hodgkin's; NHL; B-Cell; Indolent
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma | interventions — Bortezomib; Rituximab

INTERVENTIONS:
Drug: VELCADE and rituximab

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of VELCADE when given in combination with rituximab in patients with Relapsed or Refractory Indolent B-Cell Lymphoma. This study will investigate if treatment with VELCADE and rituximab increases the time it takes your lymphoma to get worse.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject 18 years or older
* Diagnosis of B-cell lymphoma (CD20+) of

  * follicular lymphoma (grades 1, 2, and 3) or
  * marginal zone lymphoma (extranodal, nodal, and splenic)
* Documented relapse or progression following prior anti-neoplastic treatment.
* At least 1 measurable lymph node mass that is >1.5 cm.
* No active CNS lymphoma
* Voluntary consent

Exclusion Criteria:

* Previous treatment with VELCADE
* Any anti-neoplastic or experimental therapy within 3 weeks before the first dose of study drug.
* Any treatment with nitrosoureas within 6 weeks before the first dose of study drug.
* Treatment with Zevalin™ or Bexxar® within 10 weeks before the first dose of study drug.
* Rituximab, Campath® or other unconjugated therapeutic antibody within 4 weeks before the first dose of study drug.
* Radiation therapy within 3 weeks before the first dose of study drug.
* Major surgery within 2 weeks before the first dose of study drug.
* Peripheral neuropathy or neuropathic pain
* History of allergic reaction attributable to compounds containing boron or mannitol
* Known anaphylaxis or hypersensitivity to any component of rituximab
* Diagnosed or treated for a selected malignancies other than NHL within 5 years.
* Active systemic infection requiring treatment
* Female subjects must not be pregnant, breast-feeding, or become pregnant during the course of the study.
* Male subjects who do not agree to use an acceptable method of contraception for the duration of the study
* Any serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Concurrent treatment with another investigational agent. Concurrent participation in non-treatment studies is allowed, if it will not interfere with participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66
Dates: Start 2004-05; Primary Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - UCLA School of Medicine, Los Angeles, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Emory University Cancer Institute, Winship Cancer Institute, Atlanta, Georgia
  - Georgia Cancer Specialists, Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Midwest Cancer Research Group, Skokie, Illinois
  - Cancer Center of Kansas, Wichita, Kansas
  - Oncology/Henmatology Associates of Kansas City, Kansas City, Missouri
  - Mid Ohio Oncology/Hematology Inc., Columbus, Ohio
  - Charleston Cancer Center, Charleston, South Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
  - FNVHO - US Oncology, Fairfax, Virginia